CLINICAL TRIAL: NCT04355065
Title: Randomized Study of Personalized Cognitive Training With Virtual Reality Technology (The Secret Trail of Moon) Versus Online Therapeutic Chess Cognitive Training Versus Usual Treatment (TAU) in Attention Deficit Hyperactivity Disorder (ADHD):a Clinical Trial"
Brief Title: The Secret Trail of Moon (Serious Videogame) and Chess on ADHD: a Clinal Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Ministerio de Economía y Competitividad, Spain (Other Government); Gammera Nest Technology Company (Unknown)
Responsible Party: Principal Investigator, Dr. Hilario Manuel Blasco Fontecilla, Psychiatrist, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hilario Blasco Fontecilla
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention deficit hyperactivity disorder; Serious videogames; Cognitive training; Chess
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study is prospective, unicentric, ramdominated, superiority with a control group and with a sample of 105 patients diagnosed with ADHD and pharmacologically stable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Training with Virtual Reality Videogame (Experimental): The Secret trail of mon is a therapeutic video game that has been created for the cognitive training of patients with ADHD.
  Five mechanisms have been designed to work on five cognitive functions that are deficient in ADHD: attention, memory, reasoning, planning and visuospatial ability.
  Patients have to go to the hospital once a week for training sessions of approximately forty minutes duration during 12 weeks.
  Interventions: Behavioral: Cognitive Traning with The Secret Trail of Moon
- Cognitive Training with Therapeutic chess (Experimental): The training in Therapeutic chess consists of four sections:
  Video tutorial: Weekly videos have been recorded in which a chess board and the image of the psychologist explaining the lesson appear. Each week a chess concept will be explained.
  Traditional chess exercises Therapeutic chess exercises: The exercises use the elements of chess but it is not necessary to know how to play chess to perform them. The purpose of the exercise is to work on a specific cognitive area each week.
  Playing online games: The patient must play a minimum of 2 online games on the chess platform chess24.es . The psychologist will follow the progress of each patient.
  At the end of the week, the patient should send an email to the psychologist with the completed exercises and then they will receive a personalised email. This group carries out all the treatment online from their home.
  Interventions: Behavioral: Cognitive Traning with Therapeutic Chess
- Control Group (Active Comparator): This group corresponds to the control group. The control group continues with their prescribed pharmacological treatment without any cognitive intervention. The participants of this group are contacted by telephone once a week to follow up on possible difficulties and/or side effects.
  Interventions: Drug: Control Group

INTERVENTIONS:
Behavioral: Cognitive Traning with The Secret Trail of Moon — Patients are pharmacologically stable and receive a cognitive intervention with our videogame once a week in the hospital.
  Arms: Cognitive Training with Virtual Reality Videogame
Behavioral: Cognitive Traning with Therapeutic Chess — This group is pharmacologically stable. This group performs cognitive training through a therapeutic chess protocol designed by a chess psychologist. The training is done from home and we contact them weekly to correct the exercises done and to follow up.
  Arms: Cognitive Training with Therapeutic chess
Drug: Control Group — These patients continue their stable pharmacological treatment and do not receive any additional cognitive intervention.
  They are contacted weekly by phone to follow up on the group.
  Arms: Control Group

SUMMARY:
Blackground:

Currently research on alternative forms of cognitive training in patients diagnosed with ADHD is gaining interest. Especially, the use of Virtual Reality video games. Our team has developed an innovative video game based on Virtual Reality, "The Secret Trail of Moon (TSTM) as a cognitive tool to train 5 main areas of deficit in patients with ADHD. It is superiority study comparing TSTM with therapeutic chess and control group.

Methods:

This study is prospective, unicentric, randomized with a control group. 105 patients diagnosed with ADHD and pharmacologically stable, aged between 12 and 22 years. These patients will be randomized intro three groups: TSTM group (The Secret Trail of Moon); TC group (Therapeutic Chess) and CG (Control Group). Objective and subjective measures of the patient, parents and teachers will be included. Patients´visit will be different for each group. The TSTM group will have 15 face-to face visits: pre-inclusion visit, inclusion visit, 12 training visits and final visit. CT and GC group patients will have 3 face-to- face visits (pre-inclusion, initial visit and final visit) and 12 email or phone communications during training.

Discussion: This study aims to demonstrate the added efficacy of cognitive training to drug treatment. It is a study that tries to demonstrate the superiority of cognitive training with TSTM compared to a traditional cognitive training (TC) and a control group.

TSTM is presented as a new and powerful cognitive tool thanks to four factors that make it unique: the feeling of immersion in the scenarios, the variety of mechanics, the personalization and the playful aspect.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults (male and female) between the ages of 12 and 22.
* Diagnosis of Attention Deficit Hyperactivity Disorder.
* Patients with stable pharmacological treatment for ADHD.
* Signature of the informed consent by the patient and their parents.

Exclusion Criteria:

* A diagnosis of ADHD comorbid with autism spectrum disorder or mental retardation.
* Suffering from epilepsy.
* Mobility plans in the next 3 months.
* Plans to begin other psychological treatment, including cognitive-behavioral psychotherapy in the next 3 months.
* Possibility of suicide risk as assessed by the clinician.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-01-22 (Estimated)

PRIMARY OUTCOMES:
Behavior rating inventory executive function (BRIEF-2) | 3 months
  The BRIEF-2 is a questionnaire designed for the evaluation of executive functions in children and adolescents. It is made up of 63 items with three answer options (never, sometimes and frequently). Its correction provides four general indexes: emotional regulation, cognitive regulation, behavioral regulation and global index of executive function.

SECONDARY OUTCOMES:
Attention-Deficit Hyperactivity Disorder Rating Scale-5 (ADHD-5) | 3 months
  This scale is made up of the 18 symptoms. The symptoms are divided into 9 for inattention, 6 for hyperactivity and 3 for impulsivity. Parents and teachers must answer yes/no to each of them. For its diagnosis, 6 or more of the attention deficit symptoms and/or 6 more of hyperactivity-impulsivity symptoms must be fulfilled. Depending on the symptoms met, the inattentive, hyperactive-impulsive or combined profile is specified.
Teacher and Parent Rating Scale( SNAP-IV) | 3 months
  The SNAPIV is a scale for the assessment of ADHD symptoms. It consists of 18 scalar items from 0 to 3, of which 9 assess attention deficit and another 9 assess hyperactive-impulsive component. The cut-off points for attention deficit are 2.56 for teachers and 1.78 for parents. For hyperactivity-impulsivity they are 1.78 for teachers and 1.44 for parents. For both components, the points are 2 for teacher and 1.67 for parents.
The Conners Comprehensive Behaviour Rating Scale (CBRS) | 3 months
  The Conners scales are a set of scales for the assessment of patients with ADHD. This revised and abbreviated version of the Conners scale is designed to be answered by parents of children ages 6-18. It consists of 10 items with a Likert type response: 0= not true at all/never; 1= just a little true/occasionally; 2= Pretty much true/often; 3=very much true/very often.
  The cut-off points are divided by gender. For children, a score above 16 is suspected ADHD. While for girls, a suspected diagnosis of ADHD is from 12 points
Emotional Quotient Inventory: Youth Version.(BarOn EQ-i:YV) | 3 months
  The BarOn is a questionnaire that it has 60-question, answered by children and young people from 7 to 18 years old. It provides information on total emotional intelligence, divided into four subscales: intrapersonal, interpersonal, stress management and adaptability. It also provides a general mood scale and other validation scales such as positive impression and inconsistency.
TEA Questionnaire for the Evaluation of ADHD and Executive Functions (ATENTO) | 3 months
  The ATENTO is a questionnaire in the process of validation that give a complete profile of the clinical symptoms of ADHD. This questionnaire has three parts: the first, with 125 items is common to all ages from 3 to 18 years. The second part, with 40 items had to be filled in if it was a patient from 3 to 6 years old and was not used in our study since the sample started from 7 years old. The third and last part, with 48 items, evaluated the population from 6 to 18 years old. All the items are of the likert type, and the parents can give scores of: 1= never or almost neves; 2= Rarely; 3= Sometimes; 4= Many times; 5= Always or almost always.
Conners Continuous Performance Test 3rd Edition (CPT-3) | 3 months
  The Conners CPT-3 is a computerized, standardized, and validated application test for different age and gender groups. The test consists of pressing a button each time a letter (target) appears on the screen, except for the letter X (non-target), which should not be pressed. The duration is approximately 14 minutes and the presentation interval between letters is variable (1, 2 and 4 seconds). The test provides results on hits, error of omission (undetected target) and errors of commission (reacted non-target), which are considered a measure of impulsivity. In addition, CPT3-3 provides information on mean reaction time and reaction time variability of hits.
Udvalg für Kliniske Undersolgelser (UKU) | 3 months
  The UKU is a tool designed to evaluate possible secondary symptoms that happen during the week. This scale is not included in the assessment phases. Only the TSTM group should complete the scale after each cognitive training session.

CONTACTS AND LOCATIONS:
Locations (1):
- Puerta de Hierro University Hospital, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Blasco-Fontecilla H, Gonzalez-Perez M, Garcia-Lopez R, Poza-Cano B, Perez-Moreno MR, de Leon-Martinez V, Otero-Perez J. Efficacy of chess training for the treatment of ADHD: A prospective, open label study. Rev Psiquiatr Salud Ment. 2016 Jan-Mar;9(1):13-21. doi: 10.1016/j.rpsm.2015.02.003. Epub 2015 Apr 22. English, Spanish. PMID 25911280
- [Result] Bul KC, Franken IH, Van der Oord S, Kato PM, Danckaerts M, Vreeke LJ, Willems A, van Oers HJ, van den Heuvel R, van Slagmaat R, Maras A. Development and User Satisfaction of "Plan-It Commander," a Serious Game for Children with ADHD. Games Health J. 2015 Dec;4(6):502-12. doi: 10.1089/g4h.2015.0021. Epub 2015 Sep 1. PMID 26325247
- [Result] Bashiri A, Ghazisaeedi M, Shahmoradi L. The opportunities of virtual reality in the rehabilitation of children with attention deficit hyperactivity disorder: a literature review. Korean J Pediatr. 2017 Nov;60(11):337-343. doi: 10.3345/kjp.2017.60.11.337. Epub 2017 Nov 27. PMID 29234356
- [Result] Barkley RA. Behavioral inhibition, sustained attention, and executive functions: constructing a unifying theory of ADHD. Psychol Bull. 1997 Jan;121(1):65-94. doi: 10.1037/0033-2909.121.1.65. PMID 9000892
- [Result] Brown M, O'Neill N, van Woerden H, Eslambolchilar P, Jones M, John A. Gamification and Adherence to Web-Based Mental Health Interventions: A Systematic Review. JMIR Ment Health. 2016 Aug 24;3(3):e39. doi: 10.2196/mental.5710. PMID 27558893
- [Result] Lau HM, Smit JH, Fleming TM, Riper H. Serious Games for Mental Health: Are They Accessible, Feasible, and Effective? A Systematic Review and Meta-analysis. Front Psychiatry. 2017 Jan 18;7:209. doi: 10.3389/fpsyt.2016.00209. eCollection 2016. PMID 28149281
- [Derived] Rodrigo-Yanguas M, Martin-Moratinos M, Gonzalez-Tardon C, Sanchez-Sanchez F, Royuela A, Bella-Fernandez M, Blasco-Fontecilla H. Effectiveness of a Personalized, Chess-Based Training Serious Video Game in the Treatment of Adolescents and Young Adults With Attention-Deficit/Hyperactivity Disorder: Randomized Controlled Trial. JMIR Serious Games. 2023 Apr 24;11:e39874. doi: 10.2196/39874. PMID 37093628
- [Derived] Rodrigo-Yanguas M, Martin-Moratinos M, Menendez-Garcia A, Gonzalez-Tardon C, Royuela A, Blasco-Fontecilla H. A Virtual Reality Game (The Secret Trail of Moon) for Treating Attention-Deficit/Hyperactivity Disorder: Development and Usability Study. JMIR Serious Games. 2021 Sep 1;9(3):e26824. doi: 10.2196/26824. PMID 34468332
- [Derived] Rodrigo-Yanguas M, Martin-Moratinos M, Menendez-Garcia A, Gonzalez-Tardon C, Sanchez-Sanchez F, Royuela A, Blasco-Fontecilla H. A Virtual Reality Serious Videogame Versus Online Chess Augmentation in Patients with Attention Deficit Hyperactivity Disorder: A Randomized Clinical Trial. Games Health J. 2021 Aug;10(4):283-292. doi: 10.1089/g4h.2021.0073. PMID 34370610